CLINICAL TRIAL: NCT03693079
Title: Investigation of Wet Cupping Therapy on Heavy Metal Levels of Steel Industry Workers: A Self Controlled Interventional Study
Brief Title: Investigation of Wet Cupping Therapy on Heavy Metal Levels of Steel Industry Workers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Karabuk University (Other)
Responsible Party: Principal Investigator, SULEYMAN ERSOY, Assist.Prof. Department of Family Medicine, Karabuk University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: KBU-BAP-17/1-KA-071
Record Dates: First submitted 2018-09-30; First posted 2018-10-02 (Actual); Last update posted 2018-10-02 (Actual); Status verified 2018-07

CONDITIONS: Heavy Metal Toxicity
Keywords: heavy metal; wet cupping therapy; steel industry worker
MeSH Terms: conditions — Heavy Metal Poisoning

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Wet Cupping (Experimental): wet cupping therapy will be applied to all participants
  Interventions: Procedure: Wet cupping therapy

INTERVENTIONS:
Procedure: Wet cupping therapy — CT was applied using plastic disposable vacuum cups on the back in the 5 areas of C7 cervical spine (DU14 acupoint), T2-4 lateral spine bilaterally (BL41-42 acupoint) and T6-8 lateral spine bilaterally (BL44-46). The cupping technique procedure was conducted in five phases:
  1. Primary suction; cups are left attached to the skin for 5 minutes.
  2. Area disinfection; areas are wiped with sterile gauze after disinfection with povidone iodine.
  3. Scarification; Superficial incisions (20-30 gauge), 5 mm length and 1-2 mm depth, are made on the skin with a sterile, number 11 surgical blade.
  4. Bloodletting and secondary suction; the cups which had been previously removed are placed again on the scarified areas Blood leaks from the capillary vessels of the skin and subcutaneous tissue and fills the cups, which are left in place for 15 minutes.
  5. Removing and dressing; the cups full of blood are removed. The areas of application are wiped with sterile gauze and then a dressing is applied

SUMMARY:
This interventional study investigates the efficacy of Wet cupping therapy on heavy metal levels.The levels of the selected heavy metals will be measured in the blood samples obtained from the participants before and after the interventions

DETAILED DESCRIPTION:
Wet cupping therapy (WCT) is a traditional therapy which was used for centuries especially for detoxifiying purposes.Current literature also points out its blood clarifiying capacity in order to illuminate the underlying mechanism of this ancient treatment.

Steel industry workers, different from the general population are exposed to heavy metals more often.Conducting a study in this special group where we will evaluate the levels of selected heavy metals in blood before and after the three sessions of WCT might let us know its detoxifiying capacity based on measurable parameters.

ELIGIBILITY:
Inclusion Criteria:

* Healthy individuals
* Iron and Steel industry workers

Exclusion Criteria:

* having any chronic disorder
* being on daily medication
* wet cupping application in the last 6 months

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 44 (Actual)
Dates: Start 2017-09-03 (Actual); Primary Completion 2018-08-01 (Actual); Study Completion 2018-10-01 (Actual)

PRIMARY OUTCOMES:
Levels of the selected heavy metals in venous blood samples before and after the interventions | 3 months
  the levels of the calculated heavy metals will be in ppm

SECONDARY OUTCOMES:
Levels of the selected heavy metals in cupping blood samples obtained during the first intervention | 1 month
  the levels of the calculated heavy metals will be in ppm

CONTACTS AND LOCATIONS:
Locations (1):
- Suleyman Ersoy, Safranbolu, Karabük Province, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided